CLINICAL TRIAL: NCT04521764
Title: Phase I Trial of Intratumoral Administration of a Measles Virus Derivative Expressing the Helicobacter Pylori Neutrophil-Activating Protein (NAP) (MV-s-NAP) in Patients With Metastatic Breast Cancer
Brief Title: A Vaccine (MV-s-NAP) for the Treatment of Patients With Invasive Metastatic Breast Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MC1733; NCI-2020-06009 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 17-008299 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2020-08-17; First posted 2020-08-21 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Anatomic Stage IV Breast Cancer AJCC v8; Invasive Breast Carcinoma; Metastatic Breast Adenocarcinoma; Recurrent Breast Carcinoma; Stage IV Breast Cancer AJCC v6 and v7
MeSH Terms: conditions — Breast Neoplasms | interventions — Magnetic Resonance Spectroscopy; X-Rays; Biopsy; Specimen Handling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (single treatment MV-s-NAP) (Experimental): Patients receive MV-s-NAP IT on day 1 in the absence of disease progression or unacceptable toxicity. Patients undergo CT scan, MRI, tumor biopsy, and blood and urine sample collection throughout the study.
  Interventions: Biological: Oncolytic Measles Virus Encoding Helicobacter pylori Neutrophil-activating Protein; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Biopsy; Procedure: Biospecimen Collection
- Cohort 2 (Every 21 day MV-s-NAP) (Experimental): Patients receive MV-s-NAP IT on day 1 of each cycle. Cycles repeat every 21 days for up to 3 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo CT scan, MRI, tumor biopsy, and blood and urine sample collection throughout the study. (CLOSED TO ACCRUAL 6/9/2025)
  Interventions: Biological: Oncolytic Measles Virus Encoding Helicobacter pylori Neutrophil-activating Protein; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Biospecimen Collection
- Cohort 3 (Every 14 day MV-s-NAP) (Experimental): Patients receive MV-s-NAP IT on day 1 of each cycle. Cycles repeat every 14 days for up to 3 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo CT scan, MRI, tumor biopsy and blood and urine sample collection throughout the study.
  Interventions: Biological: Oncolytic Measles Virus Encoding Helicobacter pylori Neutrophil-activating Protein; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Biopsy; Procedure: Biospecimen Collection

INTERVENTIONS:
Biological: Oncolytic Measles Virus Encoding Helicobacter pylori Neutrophil-activating Protein — Given IT
  Other Names: MV Encoding NAP; MV-s-NAP; Oncolytic Measles Virus Encoding H. pylori NAP
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT scan; Computed Axial Tomography; computerized axial tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT SCAN; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Magnetic Resonance / Nuclear Magnetic Resonance; Medical Imaging; MR; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; nuclear magnetic resonance imaging; sMRI; Structural MRI
Procedure: Biopsy — Undergo tumor biopsy
  Other Names: BIOPSY_TYPE; Bx
  Arms: Cohort 1 (single treatment MV-s-NAP); Cohort 3 (Every 14 day MV-s-NAP)
Procedure: Biospecimen Collection — Undergo blood and urine sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection

SUMMARY:
This phase I trial investigates the side effects and best dose of using a modified measles virus, MV-s-NAP, in treating patients with invasive breast cancer that has spread to other places in the body (metastatic). Both the unmodified vaccination measles virus (MV-Edm) and this modified virus (MV-s-NAP) have been shown to multiply in and destroy breast cancer cells in the test tube and in research mice. MV-s-NAP has been altered by having an extra gene (piece of deoxyribonucleic acid [DNA]) so that virus can make a protein called helicobacter pylori neutrophil activating protein (NAP) which is normally expressed in inflammatory reactions. Monitoring blood, urine, tissue, and throat swab samples, and using imaging tests may help to determine whether MV-s-NAP has any impact on the amount of disease present in metastatic breast cancer patients.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximally tolerated dose (MTD) of intratumoral administration of an Edmonston strain measles virus genetically engineered to express NAP (oncolytic measles virus encoding helicobacter pylori neutrophil-activating protein (modified virus strain neutrophil activating protein [MV-s- NAP) in patients with metastatic breast cancer.

II. To determine the safety and toxicity of one-time intratumoral administration of MV-s-NAP in patients with metastatic breast cancer.

III. To determine the safety and toxicity of serial intratumoral administration of MV-s-NAP in patients with metastatic breast cancer.

SECONDARY OBJECTIVES:

I. To assess in a preliminary fashion antitumor efficacy of this approach by following radiographic response and time to progression.

Ia. Response at and away from the site of MV-s-NAP administration will be evaluated.

CORRELATIVE OBJECTIVES:

I. To assess viremia, viral replication, and measles virus shedding/persistence following intratumoral administration.

II. To determine the time course of viral infection and viral gene expression in treated/untreated lesions.

III. To determine immune response development against MV, the therapeutic s-NAP transgene, and the tumor.

IV. To obtain preliminary assessments of PD-L1 expression in tumor cells and tumor infiltrating lymphocytes (TILs).

OUTLINE: Patients are assigned to 1 of 3 cohorts.

COHORT 1: Patients receive MV-s-NAP intratumorally (IT) on day 1 in the absence of disease progression or unacceptable toxicity. Patients undergo computed tomography (CT) scan, magnetic resonance imaging (MRI), tumor biopsy and blood and urine sample collection throughout the study.

COHORT 2 (CLOSED TO ACCRUAL 6/9/2025): Patients receive MV-s-NAP IT on day 1 of each cycle. Cycles repeat every 21 days for up to 3 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo CT scan, MRI, tumor biopsy and blood and urine sample collection throughout the study.

COHORT 3: Patients receive MV-s-NAP IT on day 1 of each cycle. Cycles repeat every 14 days for up to 3 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo CT scan, MRI, tumor biopsy and blood and urine sample collection throughout the study.

After completion of study treatment, patients are followed up every 3 months during year 1, and then every 6 months during year 2.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* COHORT 1 ONLY: Pathologically confirmed invasive breast adenocarcinoma with documented estrogen receptor (ER)/progesterone receptor (PR) /HER2 status and radiographic evidence of distant metastatic disease
* COHORTS 2 & 3 ONLY: Pathologically confirmed invasive breast adenocarcinoma with documented ER/PR/HER2 status and radiographic evidence of distant metastatic or recurrent disease
* COHORT 1 ONLY: Radiographic evidence of distant metastatic disease (using 7th edition American Joint Committee on Cancer [AJCC] criteria) with two discrete sites of measurable disease
* COHORTS 2 & 3 ONLY: Radiographic evidence of distant metastatic or recurrent disease (using 8th edition AJCC criteria) with at least one site of measurable disease
* Prior therapies:

  * Patients with ER/PR positive, HER2 negative breast cancer must have progressed through at least one prior cytotoxic regimen for advanced disease and no longer be candidates for standard endocrine therapy or combination of endocrine therapy with other agents such as CDK4/6 inhibitors
  * Patients with HER2 positive breast cancer irrespective of ER/PR status must have received or no longer be candidates for HER2 directed therapy with trastuzumab or pertuzumab
  * Patients with ER/PR/HER2 negative breast cancer must have progressed through at least one prior cytotoxic regimen for advanced disease
* COHORT 1: At least one site of recurrent/metastatic disease that measures > 1 cm in greatest dimension (> 2 cm for lung lesions) and is amenable to safe percutaneous intratumoral administration of MV-s-NAP as determined by an interventional radiologist
* COHORTS 2 & 3 ONLY: At least 1 site of recurrent/metastatic disease measuring > 1 cm in greatest dimension [> 2 cm for lung lesions] (Note that if the lesion injected in cycle 1 is not amenable to re-injection, another lesion could be selected for injection
* Absolute neutrophil count (ANC) >= 1500/uL (=< 7 days prior to registration)
* Platelets (PLT >= 100,000/uL) (=< 7 days prior to registration)
* Total bilirubin =< institutional upper limit of normal (=< 7 days prior to registration)
* Aspartate aminotransferase (AST) =< 2 x upper limit of normal (ULN) (=< 7 days prior to registration)
* Creatinine =< 1.5 x ULN (=< 7 days prior to registration)
* Hemoglobin >= 9.0 g/dL (=< 7 days prior to registration)
* Negative pregnancy test done =< 7 days prior to registration (for women of childbearing potential only)
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1 or 2
* Ability to provide informed written consent
* Willingness to return to the Mayo Clinic enrolling institution for follow-up
* Willingness to provide biologic samples for correlative research purposes
* Life expectancy >= 12 weeks
* Concomitant administration of a bone modifying agent (e.g., zoledronic acid or denosumab) is permitted for the prevention or management of skeletal related events in patients with bone metastases and documentation of tolerability with prior exposures

Exclusion Criteria:

* Known standard therapy for the patient's disease that is potentially curative or definitely capable of extending life expectancy
* Clinical or radiographic suspicion of impending visceral crisis due to invasion or compression by tumor
* Active infection =< 5 days prior to registration
* History of other malignancy =< 5 years except for non-melanoma skin cancer or carcinoma in situ of the cervix
* Any of the following prior therapies:

  * Chemotherapy =< 3 weeks prior to registration
  * Immunotherapy =< 4 weeks prior to registration
  * HER2 directed therapy =< 3 weeks prior to registration
  * Targeted therapy =< 2 weeks prior to registration (e.g., CDK4/6 inhibitors, everolimus)
  * Investigational agent =< 4 weeks prior to registration
  * Any viral or gene therapy prior to registration
* Failure to fully recover from acute, reversible effects of prior systemic therapy regardless of interval since last treatment
* New York Heart Association classification III or IV, known symptomatic coronary artery disease, or symptoms of coronary artery disease on systems review, or known cardiac arrhythmias (atrial fibrillation or supraventricular tachycardia [SVT])
* Untreated or progressive central nervous system (CNS) metastases

  * NOTE: Patients with a history of treated brain metastases (surgical resection, whole brain radiation, and/or stereotactic radiosurgery) are eligible only if they are asymptomatic and have stable MRI scans for 3 consecutive months, including < 28 days of study entry
* Standing requirement for blood product support
* Human immunodeficiency virus (HIV) positive test result or history of other immunodeficiency
* History of organ transplantation
* History of chronic hepatitis B or C
* Other concurrent chemotherapy, immunotherapy, radiotherapy, or any ancillary therapy considered investigational (utilized for a non-Food and Drug Administration [FDA]-approved indication and in the context of a research investigation)
* Any concurrent medications that the principal investigator determines could interfere with the trial
* Treatment with oral/systemic corticosteroids, with the exception of topical or inhaled steroids
* Exposure to household contacts =< 15 months old or household contact with known immunodeficiency
* Allergy to measles vaccine or history of severe reaction to prior measles vaccination
* History of receiving the measles vaccination with the "killed vaccine" between 1963-1967 without subsequent re-immunization (2 doses) with the active, live vaccination."

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2020-09-23 (Actual); Primary Completion 2027-08-15 (Estimated); Study Completion 2027-08-15 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose | During the first cycle of treatment (each cycle = 21 days)
  This is defined as the highest dose level among those under consideration where at most one of 6 patients develops a dose limiting toxicity, and two or more of the 3-6 patients treated at the next higher dose level develop a dose limiting toxicity.
Best tumor response | Up to 2 years
  The best tumor response in the injected and non-injected lesion will be determined using Response Evaluation Criteria in Solid Tumors (RECIST) criteria. Results will be tabulated for the entire cohort and by breast cancer subtype in terms of whether there was response in none of the lesions, only the injected lesion, or both lesions.
Incidence of adverse events | Up to 2 years
  The maximum grade of each type of toxicity will be recorded for each patient. For each toxicity reported by dose level, the percentage of patients developing any degree of that toxicity, as well as the percentage of patients developing a severe (grade 3 or higher) toxicity, will be determined.
Measles virus viremia | Up to 2 years
  Defined as detection of any titer of virus by quantitative real time-polymerase chain reaction performed with patient peripheral blood mononuclear cells. Viremia will be examined in terms of the day and dose level it was detected, as well as the time to recovery.
Peripheral immune response | Up to 2 years
  Peripheral immune response specific to measles virus is defined as detection of serum IgG anti-measles antibody levels of > 20.0 EU/mL by the Enzyme Immunoassay. Peripheral anti-neutrophil activating protein (NAP) transgene response will be represented by antibody titers determined by an antigen-mediated enzyme linked immunosorbent assay against purified helicobacter pylori NAP antigen. Systemic induction of HMGB1 will also be determined. All of these factors will be examined in terms of the day and dose level they were detected, as well as the time to recovery. For each dose level, the point at which viral replication and measles virus shedding is no longer seen will be tabulated.

SECONDARY OUTCOMES:
Tumor response | Up to 2 years
  The best tumor response in the injected and non-injected lesion will be determined using Response Evaluation Criteria in Solid Tumors (RECIST). Results will be tabulated by dose level and whether there was a response in none of the lesions, only the injected lesion, or both lesions.
Progression-free survival (PFS) | Up to 2 years
  PFS is defined as the time from study entry to the documentation of disease progression.
Overall survival (OS) | Up to 2 years
  OS is defined as the time from study entry to death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Siddhartha Yadav, MD, Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Viker KB, Steele MB, Iankov ID, Concilio SC, Ammayappan A, Bolon B, Jenks NJ, Goetz MP, Panagioti E, Federspiel MJ, Liu MC, Peng KW, Galanis E. Preclinical safety assessment of MV-s-NAP, a novel oncolytic measles virus strain armed with an H . pylori immunostimulatory bacterial transgene. Mol Ther Methods Clin Dev. 2022 Jul 31;26:532-546. doi: 10.1016/j.omtm.2022.07.014. eCollection 2022 Sep 8. PMID 36092362
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials